CLINICAL TRIAL: NCT06555146
Title: Glucagon-like Peptide-1's Effect on Renal Regional Blood Flow and the Renal Function in Patients With Type 2 Diabetes Mellitus
Brief Title: Semaglutide's Effect on Renal Hemodynamics and Function in Patients With Type 2 Diabetes Mellitus and Nephropathy
Acronym: Sema-RMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ali Asmar, Chief Physician, Associate Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-20036378
Record Dates: First submitted 2024-08-07; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2; Kidney Disease, Chronic
Keywords: Renal flow; Regional renal perfusion; Sodium excretion in urine; Renin angiotensin aldosterone system; Glomerular filtration rate
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — semaglutide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled crossover with around 4 weeks between study periods.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Randomized to start with Semaglutide intervention in study period 1 (Other): Placebo will be given in study period 2
  Interventions: Drug: Semaglutide, 0.5 mg/mL; Drug: Placebo, Saline
- Randomized to start with Placebo intervention in study period 1 (Other): Semaglutide will be given in study period 2
  Interventions: Drug: Semaglutide, 0.5 mg/mL; Drug: Placebo, Saline

INTERVENTIONS:
Drug: Semaglutide, 0.5 mg/mL — 1 subcutaneous injection on baseline day
Drug: Placebo, Saline — 1 subcutaneous injection on baseline day

SUMMARY:
The goal of this double-blinded, placebo-controlled, randomized, crossover study is to examine the effect of semaglutide, a glucagon-like peptide-1 receptor agonist (GLP-1RA), on renal hemodynamics and function in patients with type 2 diabetes mellitus (T2DM) and moderate chronic kidney disease (CKD).

The study will determine the effects of semaglutide on:

* Renal arterial blood flow, regional renal perfusion, and oxygenation
* Activity of the renin-angiotensin-aldosterone system (RAAS)
* The glomerular filtration rate (GFR)
* Sodium excretion in urine
* Blood pressure and heart rate

DETAILED DESCRIPTION:
Mechanistic studies conducted in healthy humans demonstrate a Glucagon-like peptide-1 (GLP-1)-mediated gut-kidney crosstalk. The expansion of extracellular fluid volume uncovers a natriuretic action of GLP-1. This feed-forward natriuretic system is associated with high renal extraction of GLP-1, suppression in circulating angiotensin II levels, and increased renal medullary and cortical perfusion and oxygenation. Besides potent glucose-lowering actions, Glucagon-like peptide-1 receptor agonists (GLP-1RAs) improve body weight, blood pressure, and dyslipidemia, and cardiovascular and renal outcome trials demonstrate beneficial actions of GLP-1RAs used in patients with type 2 diabetes mellitus (T2DM).

Thus the beneficial cardiovascular effects of GLP-1 may partly be related to renoprotection and might represent the restoration of the gut-kidney crosstalk.

The aim of the present study is to investigate possible mechanisms behind the renal effects of semaglutide in patients with type 2 diabetes mellitus and moderate chronic kidney disease.

This is a double-blinded, placebo-controlled, crossover study and patients will participate in two independent and randomized study periods with a washout period of around 4 weeks in between.

Fifteen male participants with type 2 diabetes mellitus in the age group 20-60 years are screened, randomized, and expected to complete the present study. Informed consent is obtained before the screening meeting followed by a 30-day run-in period prior to study days.

The two study periods each extend over 8 days, where all participants consume a controlled diet with fixed salt intake corresponding to a daily intake of 50-70 mmol + 2 mmol/kg sodium for 7 days. On the fourth day before each of the two baseline trials, 24-hour urine collection will be performed. Throughout the 7 days, water intake will be ad libitum and physical activity will not be allowed.

Each period consists of Baseline day (day 5) and Intervention day (day 8)

Renal flow, perfusion, and oxygenation are measured on both days, using multiparametric MRI.

Glomerular filtration rate (GFR) is measured, using Tc99m-Diethylenetriamine pentaacetic acid (DTPA) plasma clearance.

After conducting the baseline study, the participant is given a subcutaneous injection of either semaglutide or placebo.

During the intervention study, MRI is followed by catheterization of a renal vein via the femoral vein (the Seldinger technique) for blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus diagnosed through either HbA1c ≥6,5% but ≤8,5%, or <6,5% combined with either fasting plasma glucose ≥7,0 mmol/L or plasma glucose ≥11,1 mmol/L two hours after an oral glucose tolerance test (OGTT).
* Estimated glomerular filtration rate (eGFR, CKD-EPI) between 30-60 mL/min/1.73m2
* Urine Albumin:Creatinine ratio (UACR) ≥30mg/g
* Stable RAAS blockade (ACE inhibitors or angiotensin II receptor blocker (ARB) with stable dosis for 4 weeks prior to screening)
* Discontinuation of treatment with selective sodium glucose transporter inhibitors (SGLT2i), dipeptidyl peptidase 4 inhibitors (DPP-4i), GLP-1R analogs, rapid-acting and mix insulin 30 days before screening.

Exclusion Criteria:

* Immunosuppressive therapy within 30 days of screening
* Alcohol abuse
* Medical treatment with glucocorticoids
* Kidney transplantation
* Treatment for renal failure with dialysis
* Myocardial infarction within 3 months of screening
* Heart failure (NYHA 3-4)
* Dysregulated arterial hypertension (systolic blood pressure ≥180 mm Hg or diastolic blood pressure ≥ 100 mm Hg)
* Liver disease (ALAT >2 x normal value)
* Conditions which may interfere with the glucose metabolism according to the PI
* Severe claustrophobia
* Elements incompatible with MRI
* Abnormal kidney size and/or position
* Venous and arterial anatomy hindering catheterization.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Total blood flow | Measured during 30 minutes of MRI. One measurement will be done on each study day, a total of 4 measurements for each participant, over the span of the study (approximately 1 year).
  Volume of blood per unit time, ml/min
Regional renal perfusion | Measured during 30 minutes of MRI. One measurement will be done on each study day, a total of 4 measurements for each participant, over the span of the study (approximately 1 year)
  volume of blood per unit time per unit tissue mass, ml/min/g

SECONDARY OUTCOMES:
Glomerular filtration rate | Measured with Tec99-DTPA clearance. One measurement will be done on each study day, a total of 4 measurements for each participant, over the span of the study (approximately 1 year)
  Volume per unit time, ml/min
Sodium excretion in urine | One measurement will be done on each intervention day, a total of 2 measurements for each participant, over the span of the study (approximately 1 year)
  Concentration, mmol/l
Activation of the renin angiotensin aldosterone system | Blood samples will be taken 3 times on each intervention day, a total of 6 measurements for each participant, over the span of the study (approximately 1 year)
  Concentration, mmol/l
Blood pressure | Measured continuously during a 60 minute period on each intervention day, a total of 2 measurements for each participant, over the span of the study (approximately 1 year)
  mmhg
Heart Rate | Measured continuously during a 60 minute period on each intervention day, a total of 2 measurements for each participant, over the span of the study (approximately 1 year)
  Beats pr. minute

CONTACTS AND LOCATIONS:
Overall Officials: Ali Asmar, MD, PhD, Principal Investigator — Bispebjerg Hospital, Department of Clinical Physiology & Nuclear Medicine
Locations (1):
- Bispebjerg Hospital, Department of Clinical Physiology & Nuclear Medicine, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952